CLINICAL TRIAL: NCT01212874
Title: Esmolol or Nitroglycerin Infusion for Blood Pressure Control Prior to Cardiopulmonary Bypass(CPB) in Cardiac Surgery: a Randomized, Controlled Trial
Brief Title: Esmolol or Nitroglycerin Infusion for Blood Pressure Control Prior to Cardiopulmonary Bypass (CPB) in Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Richard Applegate, Principal Investigator, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5100218
Record Dates: First submitted 2010-09-23; First posted 2010-10-01 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Nitroglycerin; esmolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitroglycerin (Active Comparator): nitroglycerin titrated to control hypertension between anesthesia induction and initiation of cardiopulmonary bypass
  Interventions: Drug: nitroglycerin
- Esmolol (Active Comparator): esmolol titrated to control hypertension between anesthesia induction and initiation of cardiopulmonary bypass
  Interventions: Drug: esmolol

INTERVENTIONS:
Drug: nitroglycerin — nitroglycerin administered as an infusion following a step up/step down protocol to treat hypertension in patients undergoing cardiac surgery.
  Arms: Nitroglycerin
Drug: esmolol — esmolol will be administered by infusion following a step up / step down protocol to control hypertension.
  Arms: Esmolol

SUMMARY:
This is an investigator initiated, sponsored, open label, prospective randomized controlled trial to be performed in adult patients undergoing scheduled cardiac surgery. Patients will be randomized to esmolol infusion or nitroglycerin infusion for control of hypertension that occurs during cardiac surgery from induction of anesthesia to initiation of cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for cardiac surgery at LLUMC University Hospital will be eligible for participation in this study.

Exclusion Criteria:

1. severe LV (left ventricle)dysfunction (EF < 35%).
2. emergency procedures.
3. procedures with combined carotid artery surgery.
4. patients at high risk for stroke.
5. hemodynamically significant dysrhythmias.
6. pre-existing atrial fibrillation or high degree AV (atrioventricular block).
7. pacemaker dependency.
8. known sensitivity to beta blockers.
9. patient refusal.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Applegate II, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Esmolol | Nitroglycerin
Started | 35 | 35
Received Allocated Intervention | 13 | 12
Completed | 13 | 12
Not Completed | 22 | 23

BASELINE CHARACTERISTICS:
Groups:
- Nitroglycerin: nitroglycerin infusion titrated to control hypertension from anesthesia induction to initiation of cardiopulmonary bypass
  nitroglycerin: nitroglycerin administered as an infusion following a step up/step down protocol to treat hypertension in patients undergoing cardiac surgery.
- Esmolol: esmolol infusion titrated to control hypertension from anesthesia induction to initiation of cardiopulmonary bypass
  esmolol: esmolol will be administered by infusion following a step up / step down protocol to control hypertension.
- Total: Total of all reporting groups
Arm/Group | Nitroglycerin | Esmolol | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 19 | 42
  >=65 years | 12 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (11.6) | 61.6 (13.2) | 61.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
Body mass index kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 29.8 (5.6) | 29.5 (7.7) | 29.6 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Diastolic Blood Pressure Excursions Beyond Predetermined Lower Limits, Normalized Per Hour
Description: Area under the curve (AUC) of Diastolic Blood Pressure Excursions Beyond Predetermined Lower Limits, Normalized Per Hour from Anesthesia Induction to Initiation of Cardiopulmonary Bypass
Time Frame: Participants were followed from Anesthesia Induction to Initiation of Cardiopulmonary Bypass, an average of 5 hours
Population: Data capture failure lost data from 2 treated patients in each group; these were thus excluded from analysis.
Measure: Median (95% Confidence Interval); unit: mmHg*min/prebypass hour
Arm/Group | Esmolol | Nitroglycerin
Number analyzed (Participants) | 11 | 10
mmHg*min/prebypass hour | 97.9 [47.7 to 181.4] | 45.6 [21.0 to 93.9]
Statistical Analysis 1: Comparison: Esmolol vs Nitroglycerin; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

2. Secondary Outcome: Title: Systolic Hypertension
Description: Area under the curve (AUC) of Systolic Blood Pressure Excursions Beyond Predetermined Upper Limits, Normalized Per Hour from Anesthesia Induction to Initiation of Cardiopulmonary Bypass
Time Frame: Participants were followed from Anesthesia Induction to Initiation of Cardiopulmonary Bypass, an average of 5 hours
Population: Data capture failure lost data from 2 treated patients in each group; these were thus excluded from analysis.
Measure: Median (95% Confidence Interval); unit: mmHg*min / prebypass hour
Arm/Group | Esmolol | Nitroglycerin
Number analyzed (Participants) | 11 | 10
mmHg*min / prebypass hour | 48.6 [18.2 to 90.8] | 145.8 [79.4 to 259.9]
Statistical Analysis 1: Comparison: Esmolol vs Nitroglycerin; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Esmolol | Nitroglycerin
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
Only 25 of 70 patients received the assigned intervention. Individualized BP ranges based on day of surgery measurement likely decreased treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No